CLINICAL TRIAL: NCT02312791
Title: Observational Study of Prognosis of Inpatients Evaluated for Palliative Radiotherapy
Brief Title: Prognosis of Inpatients Evaluated for Palliative Radiotherapy
Acronym: PROGRAD
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Andre Tsin Chih Chen, MD, University of Sao Paulo
Other Study IDs: NP 683/2014
Record Dates: First submitted 2014-10-14; First posted 2014-12-09 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Cancer
Keywords: Radiation; Prognosis; Palliative Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Palliative Patients: Inpatients evaluated for palliative radiation therapy.

SUMMARY:
Understanding patient's prognosis is of utmost importance to determine radiotherapy's indication and dose/ fractionation. The investigators plan to conduct an observational study of prognosis of inpatients evaluated for palliative radiotherapy at a large cancer hospital in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* All inpatients evaluated for palliative radiation therapy at ICESP (Instituto do Cancer do Estado de Sao Paulo)

Exclusion Criteria:

* Inpatients evaluated whose intent of treatment is curative
* Patients who are unwilling to participate in the study or unwilling to sign informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients evaluated for palliative Radiation Therapy
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 9 months
  Overall Survival in the studied population

SECONDARY OUTCOMES:
Overall Survival in Each Indication of Palliative Radiotherapy | 3 months and 9 months
  Overall Survival in Each Indication of Palliative Radiotherapy.
  The indication will be as follow:
  * spinal cord compression
  * brain metastases
  * tumor bleeding
  * tumoral mass
  * Oncologic Pain
  * Superior Vena Cava Syndrome/ Airway compression
Overall Survival by Palliative Prognostic Index (PPI) | 3 months and 9 months
  Patients will be divided into 3 subgroups according to the PPI. Survival differences between the different subgroups will be compared and analyzed
Overall Survival by Survival Prognostic Score (SPS) | 3 months and 9 months
  Patients will be divided into 3 subgroups according to the SPS. Survival differences between the different subgroups will be compared and analyzed
Overall Survival by Score Index for Stereotactic Radiosurgery for Brain Metastases (SIR) | 3 months and 9 months
  Patients will brain metastases will be divided into 3 subgroups according to SIR. They will be divided into SIR 0-3; 4-7;8-10. Survival differences between the different subgroups will be compared and analyzed
Positive Predictive Value of PPI | 3 weeks and 6 weeks
  Positive Predictive Value of PPI to predict death at 3 weeks and 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Heloisa A Carvalho, MD PhD, Study Director — University of Sao Paulo; Andre T Chen, MD, Study Chair — University of Sao Paulo
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo, Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, Brazil

REFERENCES:
- [Background] Morita T, Tsunoda J, Inoue S, Chihara S. The Palliative Prognostic Index: a scoring system for survival prediction of terminally ill cancer patients. Support Care Cancer. 1999 May;7(3):128-33. doi: 10.1007/s005200050242. PMID 10335930
- [Background] Chow E, Abdolell M, Panzarella T, Harris K, Bezjak A, Warde P, Tannock I. Predictive model for survival in patients with advanced cancer. J Clin Oncol. 2008 Dec 20;26(36):5863-9. doi: 10.1200/JCO.2008.17.1363. Epub 2008 Nov 17. PMID 19018082
- [Background] Weltman E, Salvajoli JV, Brandt RA, de Morais Hanriot R, Prisco FE, Cruz JC, de Oliveira Borges S, Lagatta M, Ballas Wajsbrot D. Radiosurgery for brain metastases: who may not benefit? Int J Radiat Oncol Biol Phys. 2001 Dec 1;51(5):1320-7. doi: 10.1016/s0360-3016(01)01696-0. PMID 11728693
- [Derived] Chen ATC, Mauro GP, Gabrielli F, Chaves CLG, Castro I, Vasconcelos KM, Reis M, Saraiva T, Carvalho HA. PROGRAD - An observational study of the prognosis of inpatients evaluated for palliative radiotherapy. Radiother Oncol. 2018 May;127(2):299-303. doi: 10.1016/j.radonc.2018.03.021. Epub 2018 Apr 3. PMID 29625809